CLINICAL TRIAL: NCT07129187
Title: An Open-label, Single-arm, Multicenter Study of SHR-A1811 as Neoadjuvant Therapy in HER2-positive Breast Cancer Patients With Suboptimal Neoadjuvant Response
Brief Title: SHR-A1811 for HER2-positive Breast Cancer With Suboptimal Neoadjuvant Response
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chuan Wang (Other)
Responsible Party: Sponsor-Investigator, Chuan Wang, MD, Fujian Medical University Union Hospital
Organization: Fujian Medical University Union Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-124
Record Dates: First submitted 2025-08-01; First posted 2025-08-19 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Early Breast Cancer; HER2 + Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
Keywords: neoadjuvant therapy; antibody drug conjugate; SHR-A1811; suboptimal response
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 (Experimental)
  Interventions: Drug: SHR-A1811

INTERVENTIONS:
Drug: SHR-A1811 — Drug: SHR-A1811 4.8mg/kg

SUMMARY:
This is an open-label, single-arm, multicenter clinical study to evaluate the efficacy and safety of SHR-A1811 in early or locally advanced HER2-positive breast cancer patients with suboptimal response to neoadjuvant regimen. Patients who were determined by the researchers to have poor therapeutic effect will switch to SHR-A1811.

DETAILED DESCRIPTION:
Patients will receive SHR-A1811, until completion or treatment discontinuation due to progression, toxicity, or withdrawal. The primary endpoint is tpCR (ypT0/is ypN0). Secondary endpoints include bpCR, RCB, EFS, and safety. The study will recruit 30 eligible patients from multiple centers in China.

ELIGIBILITY:
Inclusion Criteria:

* 1.Female patients with newly diagnosed breast cancer aged 18 to 70 years old;
* 2.Early or locally advanced HER2-positive invasive breast cancer;
* 3.Known hormone receptor status;
* 4.ECOG score of 0-1;
* 5.Patients who were determined by the researchers to have poor therapeutic effect after 4 cycles of neoadjuvant therapy;
* 6.Organ function levels must meet the following requirements:
* 7.Women of childbearing age must undergo a serum pregnancy test within 7 days before enrollment, with a negative result, and be willing to use a medically approved highly effective contraceptive method during the study and within 3 months after the last administration of the study drug.
* 8.The subjects voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* 1. Patients with metastatic or bilateral breast cancer, or inflammatory breast cancer
* 2. Patients with grade 3 or higher thrombocytopenia during previous treatment, or grade 3 or higher nausea and vomiting despite primary prevention
* 3. History of other malignant tumors (except cured carcinoma in situ of the cervix, basal cell carcinoma, etc.) and related treatment history
* 4. Patients who received major non-breast cancer surgery within 4 weeks before enrollment and have not recovered (except biopsy and PICC)
* 5. Autoimmune diseases (except special cases such as hypothyroidism and stable type 1 diabetes)
* 6. Interstitial lung disease, non-infectious pneumonia, uncontrolled systemic diseases
* 7. History of or planned administration of live attenuated vaccines within 28 days
* 8. HIV infection, active hepatitis (hepatitis B, hepatitis C, etc.), autoimmune hepatitis
* 9. Severe infection within 4 weeks, CTCAE grade ≥ 2 active infection within 2 weeks (except neoplastic fever), or evidence of active tuberculosis within 1 year
* 10. History of allogeneic bone marrow or solid organ transplantation
* 11. Peripheral neuropathy of grade ≥ 2
* 12. Severe heart diseases
* 13. Receipt of systemic immunostimulant therapy within 4 weeks
* 14. Receipt of systemic immunosuppressant therapy within 2 weeks (except local or physiological dose of hormones)
* 15. Allergy to study drugs/excipients, or history of severe allergic reaction to other monoclonal antibodies
* 16. Pregnant or lactating women; fertile women with positive pregnancy test or unwilling to take effective contraception throughout the trial
* 17. History of neurological/psychiatric disorders , or history of substance abuse, alcoholism, or drug addiction
* 18. Other circumstances deemed unsuitable for enrollment by the researcher

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
tpCR | immediately after surgery
  It is defined as the absence of residual invasive carcinoma in the resected breast cancer specimens stained with hematoxylin and eosin, and no cancer metastasis in all ipsilateral lymph node samples, after completion of neoadjuvant therapy and surgery.

SECONDARY OUTCOMES:
Breast Pathological Complete Response | immediately after surgery
  It is defined as the absence of residual invasive carcinoma in the primary breast lesion after neoadjuvant therapy, with the permission of residual ductal carcinoma in situ within the primary breast lesion.
event free survival | until the end of the study
residual cancer burden | immediately after surgery